CLINICAL TRIAL: NCT02830841
Title: Remote Ischemic Preconditioning Protects Against Hepatic Ischemic and Reperfusion Injury in Pediatric Living Donor Liver Transplantation
Brief Title: Liver Protection of RIPC in Pediatric Living Donor Liver Transplantation
Acronym: RIPC-PLDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Renji[2016]002k
Record Dates: First submitted 2016-06-27; First posted 2016-07-13 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Hepatic Ischemic and Reperfusion Injury
Keywords: RIPC; hepatic ischemic and reperfusion injury; pediatric living donor liver transplantation
MeSH Terms: conditions — Reperfusion Injury

ARMS (4):
- DR-RIPC (donor and recipient RIPC group) (Experimental): Both donors and recipients receive remote ischemic preconditioning, with three 5-min cycles of remote limb ischemia, which was induced by an automated cuff-inflator placed on the right upper arm(donor) or right lower limb(recipient) and inflated to 15 mmHg above systolic pressure, with an intervening 5 min of reperfusion during which the cuff was deflated.
  Interventions: Device: remote ischemic preconditioning(RIPC)
- S-RIPC (sham RIPC) (Sham Comparator): Patients had a deflated cuff placed on the right upper arm or right lower limb for 30 min
  Interventions: Device: Sham RIPC
- R-RIPC (recipient RIPC group) (Experimental): Recipients receive remote ischemic preconditioning, with three 5-min cycles of remote limb ischemia, which was induced by an automated cuff-inflator placed on the right lower limb and inflated to 15 mmHg above systolic pressure, with an intervening 5 min of reperfusion during which the cuff was deflated.
  Interventions: Device: remote ischemic preconditioning(RIPC)
- D-RIPC (donor RIPC group) (Experimental): Donors receive remote ischemic preconditioning, with three 5-min cycles of remote limb ischemia, which was induced by an automated cuff-inflator placed on the right upper arm and inflated to 15 mmHg above systolic pressure, with an intervening 5 min of reperfusion during which the cuff was deflated.
  Interventions: Device: remote ischemic preconditioning(RIPC)

INTERVENTIONS:
Device: remote ischemic preconditioning(RIPC) — After anesthesia induction, donors or recipients will be treated with automated blood pressure cuffs on their upper arms to receive RIPC by cuff inflation (to 15mmHg above systolic pressure) for 5 minutes and left inflated for 5 minutes. The cuff will then be deflated to 0 mm Hg and left uninflated for 5 minutes. This cycle will be performed 3 times in total.
  Arms: D-RIPC (donor RIPC group); DR-RIPC (donor and recipient RIPC group); R-RIPC (recipient RIPC group)
Device: Sham RIPC — Only blood pressure cuff will be placed to the patient, but no inflation or deflation will be performed.
  Arms: S-RIPC (sham RIPC)

SUMMARY:
Remote ischemic preconditioning(RIPC) is emerging as an promising therapeutic paradigm to combat the detrimental impact of ischemic and reperfusion injury. In liver transplantation, ischemic and reperfusion injury severely impacts the post-surgery liver function and patient outcome. This prospective, double blind, randomized clinical trial is aimed to test the protective effect of RIPC against hepatic ischemic and reperfusion injury in pediatric liver transplantation.

DETAILED DESCRIPTION:
Pediatric liver transplantation remains the major therapeutic strategy for pediatric biliary atresia patients. With almost 60 years of improvements and refinements in surgical techniques and perioperative management standards, liver transplantation is gaining popularity and gradually turns out to be the only curative treatment option for patients with irrevocable liver failure, such as childhood acute or chronic liver failure, inherited liver diseases and also biliary atresia. In liver transplantation, hepatic ischemic and reperfusion injury (HIRI) remains to be a critical clinical issue. Importantly, it is well known that the severity of HIRI may have fundamental impact on the transplanted organ function and long term graft survival. Furthermore, pediatric patients are more venerable and less tolerated to receive an ischemic donor liver due to their small body weight.Although detrimental impact of HIPI on graft function has long been recognized, little progress has been made to attenuate the severity of the HIPI compared to cardiac ischemic and reperfusion (IR) injury. In experimental animal models, remote ischemic preconditioning has been consistently shown to have beneficial effects. However, this protective paradigm has yet not been tested in liver transplantation patients in clinical scenario. Considering the growing number of pediatric patients undergoing liver transplantation and their possibly underdeveloped organ function, the investigators sought to determine whether remote ischemic preconditioning could ameliorate HIPI and improve long term graft/patient survival in pediatric liver transplantation patients using this double-blind randomized clinical trial.

ELIGIBILITY:
The inclusion criteria were as follows:

1. American society of anesthesiologists score of I-III;
2. age of 3-72 months
3. elective living LT surgery.

The exclusion criteria were as follows:

1. peripheral vascular disease;
2. history of thromboembolism;
3. systemic or local infection before surgery;
4. autoimmune diseases;
5. severe congenital heart disease
6. history of LT.

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Postoperative maximum AST | Postoperative 0-7 day
  Postoperative maximum aspartate transaminase (AST)
Postoperative maximum ALT | Postoperative 0-7 day
  Postoperative maximum alanine transaminase (ALT)

SECONDARY OUTCOMES:
Occurrence of early graft dysfunction(EAD) | 7 days after surgery
  occurrence of early graft dysfunction
Number of recipients with primary nonfunction | 7 days after surgery
  Number of recipients with primary nonfunction
Number of recipients/donors with postoperative complications | 7 days after surgery
  Number of recipients/donors with postoperative complications
The overall survival of recipients | 1-year and 3-year overall survival of recipients
  1-year and 3-year overall survival of recipients after liver transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Zarbock A, Schmidt C, Van Aken H, Wempe C, Martens S, Zahn PK, Wolf B, Goebel U, Schwer CI, Rosenberger P, Haeberle H, Gorlich D, Kellum JA, Meersch M; RenalRIPC Investigators. Effect of remote ischemic preconditioning on kidney injury among high-risk patients undergoing cardiac surgery: a randomized clinical trial. JAMA. 2015 Jun 2;313(21):2133-41. doi: 10.1001/jama.2015.4189. PMID 26024502
- [Background] Bulluck H, Candilio L, Hausenloy DJ. Remote Ischemic Preconditioning: Would You Give Your Right Arm to Protect Your Kidneys? Am J Kidney Dis. 2016 Jan;67(1):16-9. doi: 10.1053/j.ajkd.2015.08.018. Epub 2015 Sep 16. No abstract available. PMID 26385818